CLINICAL TRIAL: NCT03649022
Title: "Ventricular Tachycardia Ablation Registry". Italian Registry of Substrate Mapping and VT Ablation With the Precision Mapping System and Flexability Catheter.
Brief Title: "Ventricular Tachycardia Ablation Registry".
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Paolo Della Bella (Other)
Responsible Party: Sponsor-Investigator, Paolo Della Bella, MD, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: OSR-ARITM-001
Record Dates: First submitted 2018-08-08; First posted 2018-08-28 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Catheter ablation — Ventricular Tachycardia ablation, that will be performed per clinical practice, by using EnSite Precision mapping system with the Flexability catheter (St.Jude, now Abbott)

SUMMARY:
Catheter ablation of Ventricular Tachycardias is a well-established approach in clinical practice in patients with Implantable Cardioverter Defibrillator (ICD) implanted. Previous studies have shown a significant reduction in appropriate shocks (~ 20%) and a significant reduction in hospitalizations for cardiovascular reasons (~ 12%) in patients with ischemic heart disease treated with ablation. Recent works have also shown the effectiveness of the ablation procedure using as procedural target the reduction of late potentials. However, actually it is necessary to have an homogenize and accepted mapping scheme in Sinus Rhythm to ablate Ventricular Tachycardias related to scar substrate in patients with:

* Previous MI
* Previous myocarditis
* Arrhythmogenic Right Ventricular Dysplasia (ARVD)
* Idiopathic Dilated Cardiomyopathy (IDCM)

Scope of the registry is to collect data during cardiac mapping in Sinus Rhythm in patients indicated for Ventricular Tachycardia ablation, that will be performed per clinical practice, by using the St. Jude Medical EnSiteTM PrecisionTM mapping system.

The objective of the present registry is: to assess the acute and long-term efficacy of the strategy of substrate abolition (abolishment of complex and late potentials) guided by electroanatomic mapping with Precision software.

DETAILED DESCRIPTION:
This is an Italian multicenter, observational, prospective and retrospective registry.

Data will be collected during enrollment/baseline, procedure, pre-discharge and during the follow-up visits according to the standard practice of participating centers, with mandatory visits at 6 and 12 months. Data can also be collected retrospectively, prior informed consent of the patient.

The planned enrollment duration is approximately 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an implanted ICD
* Patients with indication to Ventricular Tachycardia Ablation procedure, supported by EnSite Precision 3D mapping system (previous MI, myocarditis, ARVD, IDCM)
* Age 18 years or more
* Able to provide an informed consent to participate to the registry and available to respect the assessments described in the protocol

Exclusion Criteria:

* Contraindication to anticoagulants
* Presence of thrombi
* Presence of Mitral and Aortic prosthetic valve
* Recent (<3 months) myocardial infarction or unstable angina or Coronary Artery Bypass
* Pregnant or nursing
* Ventricular Tachycardia caused by reversible pathology
* < 1 Year life expectancy according to the investigator
* Contraindication to the use of ablation/diagnostic catheters or to cardiac catheterism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population of patients with defibrillator, indicated to perform catheter ablation of ventricular tachycardia related to substrate scar due to previous MI, previous myocarditis and arrhythmogenic right ventricular dysplasia, idiopathic dilated cardiomyopathy guided by electroanatomic mapping system.
Sampling Method: Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Late potential abolition and ventricular tachycardia noninducibility | Intraprocedural
  Combined procedural endpoint of late potential (LP) abolition and VT noninducibility (endpoint expected in 50% of cases).
  LP abolition assessed as % of persistent LP area at remap after ablation, compared to the basal activation map.
Ventricular tachycardia recurrence | 12 months
  Freedom from Ventricular Tachycardia episodes requiring ICD Intervention (shock or Anti-Tachycardia Pacing)

SECONDARY OUTCOMES:
Complications | During hospitalization: starting during the procedure until discharge
  Periprocedural complications
Complications | 12 months
  Long term catheter ablation complications
Procedural parameters | Intraprocedural
  Procedure duration measured in minutes
Procedural parameters | Intraprocedural
  Fluoroscopy exposure measured in Gycm2
Assessment of cardiac mapping system EnSite Precision™ software (St.Jude, now Abbott) | Intraprocedural
  Geometry precision, descriptive
Assessment of cardiac mapping system EnSite Precision™ software (St.Jude, now Abbott) | Intraprocedural
  Mapping accuracy, descriptive
Assessment of cardiac mapping system EnSite Precision™ software (St.Jude, now Abbott) | Intraprocedural
  System overall stability, descriptive
Assessment of cardiac mapping system EnSite Precision™ software (St.Jude, now Abbott) | Intraprocedural
  Non-recoverable shifts/drifts, descriptive

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Della Bella, MD, Principal Investigator — IRCCS S Raffaele
Locations (1):
- IRCCS San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Reddy VY, Reynolds MR, Neuzil P, Richardson AW, Taborsky M, Jongnarangsin K, Kralovec S, Sediva L, Ruskin JN, Josephson ME. Prophylactic catheter ablation for the prevention of defibrillator therapy. N Engl J Med. 2007 Dec 27;357(26):2657-65. doi: 10.1056/NEJMoa065457. PMID 18160685
- [Background] Priori SG, Blomstrom-Lundqvist C, Mazzanti A, Blom N, Borggrefe M, Camm J, Elliott PM, Fitzsimons D, Hatala R, Hindricks G, Kirchhof P, Kjeldsen K, Kuck KH, Hernandez-Madrid A, Nikolaou N, Norekval TM, Spaulding C, Van Veldhuisen DJ; ESC Scientific Document Group. 2015 ESC Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death: The Task Force for the Management of Patients with Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death of the European Society of Cardiology (ESC). Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC). Eur Heart J. 2015 Nov 1;36(41):2793-2867. doi: 10.1093/eurheartj/ehv316. Epub 2015 Aug 29. No abstract available. PMID 26320108
- [Background] Silberbauer J, Oloriz T, Maccabelli G, Tsiachris D, Baratto F, Vergara P, Mizuno H, Bisceglia C, Marzi A, Sora N, Guarracini F, Radinovic A, Cireddu M, Sala S, Gulletta S, Paglino G, Mazzone P, Trevisi N, Della Bella P. Noninducibility and late potential abolition: a novel combined prognostic procedural end point for catheter ablation of postinfarction ventricular tachycardia. Circ Arrhythm Electrophysiol. 2014 Jun;7(3):424-35. doi: 10.1161/CIRCEP.113.001239. Epub 2014 May 15. PMID 24833642
- [Background] Deo R, Albert CM. Epidemiology and genetics of sudden cardiac death. Circulation. 2012 Jan 31;125(4):620-37. doi: 10.1161/CIRCULATIONAHA.111.023838. No abstract available. PMID 22294707
- [Background] Tung R, Boyle NG, Shivkumar K. Catheter ablation of ventricular tachycardia. Circulation. 2010 Jul 20;122(3):e389-91. doi: 10.1161/CIRCULATIONAHA.110.963371. No abstract available. PMID 20644021
- [Background] Aliot EM, Stevenson WG, Almendral-Garrote JM, Bogun F, Calkins CH, Delacretaz E, Bella PD, Hindricks G, Jais P, Josephson ME, Kautzner J, Kay GN, Kuck KH, Lerman BB, Marchlinski F, Reddy V, Schalij MJ, Schilling R, Soejima K, Wilber D; European Heart Rhythm Association; European Society of Cardiology; Heart Rhythm Society. EHRA/HRS Expert Consensus on Catheter Ablation of Ventricular Arrhythmias: developed in a partnership with the European Heart Rhythm Association (EHRA), a Registered Branch of the European Society of Cardiology (ESC), and the Heart Rhythm Society (HRS); in collaboration with the American College of Cardiology (ACC) and the American Heart Association (AHA). Europace. 2009 Jun;11(6):771-817. doi: 10.1093/europace/eup098. Epub 2009 May 14. No abstract available. PMID 19443434
- [Background] Kuck KH, Schaumann A, Eckardt L, Willems S, Ventura R, Delacretaz E, Pitschner HF, Kautzner J, Schumacher B, Hansen PS; VTACH study group. Catheter ablation of stable ventricular tachycardia before defibrillator implantation in patients with coronary heart disease (VTACH): a multicentre randomised controlled trial. Lancet. 2010 Jan 2;375(9708):31-40. doi: 10.1016/S0140-6736(09)61755-4. PMID 20109864
- [Background] Themistoclakis S, Raviele A, China P, Pappone C, De Ponti R, Revishvili A, Aliot E, Kuck KH, Hoff PI, Shah D, Almendral J, Manolis AS, Chierchia GB, Oto A, Vatasescu RG, Sinkovec M, Cappato R; Atrial Fibrillation Survey Investigators. Prospective European survey on atrial fibrillation ablation: clinical characteristics of patients and ablation strategies used in different countries. J Cardiovasc Electrophysiol. 2014 Oct;25(10):1074-81. doi: 10.1111/jce.12462. Epub 2014 Jul 8. PMID 24891043
- [Derived] Radinovic A, Peretto G, Sgarito G, Cauti FM, Castro A, Narducci ML, Mantovan R, Scaglione M, Solimene F, Scopinaro A, Tondo C, Filippini G, Bianco E, Bonso A, Calzolari V, Ferraris F, Zardini M, Piacenti M, D'Angelo G, Bosica F, Della Bella P. Matching Ablation Endpoints to Long-Term Outcome: The Prospective Multicenter Italian Ventricular Tachycardia Ablation Registry. JACC Clin Electrophysiol. 2023 Jun;9(6):836-847. doi: 10.1016/j.jacep.2022.10.038. Epub 2023 Jan 18. PMID 36752462